CLINICAL TRIAL: NCT03807310
Title: The Effect of Targeted Nutrient Supplementation on Physical Activity and Healthy Related Quality of Life in COPD
Brief Title: Targeted Nutrient Supplement in COPD (NUTRECOVER-trial)
Acronym: NUTRECOVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nutricia Research (Industry)
Responsible Party: Principal Investigator, Rosanne Beijers, Principal investigator, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: METC18-011; 10.2.16.119 (Other Grant/Funding Number: The Netherlands Lung Foundation)
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; nutrient supplementation; Physical activity; Health related quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Dietary Supplements; Counseling; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Next to the 166 COPD patients that receive the nutritional supplement, a subgroup of 30 healthy controls will be included for baseline comparison of the microbiome composition. These healthy controls will not be included in the intervention arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Long-drink (Experimental): 83 COPD patients will receive:
  * Targeted nutrient supplementation (Long-drink) once daily
  * Counselling once monthly
  Interventions: Dietary Supplement: Targeted nutrient supplementation (Long-drink); Behavioral: Counselling
- Group Placebo (Placebo Comparator): 83 COPD patients will receive:
  * Isocaloric placebo supplement once daily
  * Counselling once monthly
  Interventions: Dietary Supplement: Placebo supplement; Behavioral: Counselling
- Healthy control group (No Intervention): 30 healthy controls will be included for baseline comparison of the microbiome composition. These healthy controls will only perform a subset of baseline measurements and will not be included in the intervention.

INTERVENTIONS:
Dietary Supplement: Targeted nutrient supplementation (Long-drink) — Once daily for at least 12 months
  Other Names: Nutritional supplementation; Dietary supplement; Nutritional supplement; Food supplement
  Arms: Group Long-drink
Dietary Supplement: Placebo supplement — Once daily for at least 12 months
  Other Names: Non-active supplement
  Arms: Group Placebo
Behavioral: Counselling — Counselling on healthy lifestyle (in particular physical activity, smoking cessation) and weight management by motivational interviewing
  Other Names: Motivational interviewing
  Arms: Group Long-drink; Group Placebo

SUMMARY:
The overall objective is to investigate the efficacy of targeted nutrient supplementation on daily physical activity level as well as generic health status in patients with COPD. Additionally the investigators aim to investigate the relative effect of targeted nutrient supplementation on the recovery after hospitalization for a COPD exacerbation. The secondary objective is to investigate the effect of targeted nutrient supplementation on mental health, physical performance, blood markers, patient related outcomes and gut health. Additionally, a secondary objective is to compare the gut microbiome composition of patients with COPD compared to healthy controls.

DETAILED DESCRIPTION:
Rationale: Impaired physical and mental health are common features in COPD adversely affecting disease course and quality of life. Furthermore, nutritional status is often impaired due to dietary and plasma nutrient deficiencies, decreased muscle oxidative metabolism and impaired intestinal permeability. The investigators hypothesize that targeted nutrient supplementation can lead to gut-muscle-brain axis-mediated amelioration of physical, cognitive and mental health domains, resulting in a healthier lifestyle, in patients with COPD.

Study design: Randomized, placebo-controlled, double-blind trial.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The nutrient supplement is hypothesized to have beneficial effects on general health because it applies physical and mental health domains. The healthy lifestyle counselling aims to improve medical adherence, to address a healthier lifestyle and to manage weight loss which would contribute to improved general health. Risks and inconveniences are limited to the time investment associated with taking the supplements and measuring days. During the test-days various non-invasive measurements as well as minor invasive blood sampling will be performed. The investigators expect no risk of the nutrient supplementation. Healthy controls will only attend a subgroup of baseline measurements which are limited to non-invasive measurements and one minor invasive blood sampling. Healthy controls will not receive the nutritional supplement.

ELIGIBILITY:
Inclusion Criteria COPD Patients:

* COPD patients with moderate to very severe disease stage according to GOLD criteria (i.e. GOLD stage II-IV);
* Medically stable.

Exclusion Criteria COPD Patients:

* Age <18 years;
* Allergy or intolerance to components of the study product;
* Not willing or not able to quit vitamin D or fatty acid supplement intake;
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements (e.g. leg amputation) or patients suffering from other acute or unstable chronic diseases that will compromise the study outcome (e.g. active cancer requiring treatment);
* Participation in any other study involving investigational or marketed products concomitantly or within four weeks prior to entry into the study;
* Patients with terminal illness;
* Recent hospital admission (<4 weeks prior to the start of the study);
* Temporary oral steroid or antibiotics use due to a COPD exacerbation in the last 4 weeks;
* Lung malignancy in the previous 5 years;
* Diagnosis of dementia or neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease, Huntington's chorea, frontotemporal dementia) in the medical records;
* Recent diagnosis of cerebral conditions (<1 year e.g. cerebral infarction, hemorrhage, brain tumors, transient ischemic attack) in the medical records;
* Any medical condition that significantly interferes with digestion and/or gastrointestinal function (e.g. short bowel syndrome, inflammatory bowel disease, gastric ulcers, gastritis, (gastro)-enteritis, GI-cancer) as judged by the investigator.

Inclusion Criteria Healthy Controls

* Forced expiratory volume in 1 second/Forced vital capacity > 0.7;
* Medically stable.

Exclusion Criteria Healthy Controls

* Age <18 years;
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements (e.g. leg amputation) or patients suffering from other acute or unstable chronic diseases that will compromise the study outcome (e.g. active cancer requiring treatment);
* Participation in any other study involving investigational or marketed products concomitantly or within four weeks prior to entry into the study;
* Patients with terminal illness;
* Recent hospital admission (<4 weeks prior to the start of the study);
* Temporary antibiotics use in the last 4 weeks;
* Lung malignancy in the previous 5 years;
* Diagnosis of dementia or neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease, Huntington's chorea, frontotemporal dementia) in the medical records;
* Recent diagnosis of cerebral conditions (<1 year e.g. cerebral infarction, hemorrhage, brain tumors, transient ischemic attack) in the medical records;
* Any medical condition that significantly interferes with digestion and/or gastrointestinal function (e.g. short bowel syndrome, inflammatory bowel disease, gastric ulcers, gastritis, (gastro)-enteritis, GI-cancer) as judged by the investigator.
* Diagnosis of any chronic lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity level assessed by measuring step count with accelerometry | 0, 3, and 12-14 months and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later
  Subjects will wear an activPAL accelerometer for 1 week to assess physical activity.
Change in generic health status measured by EuroQol-5 dimensions (EQ-5D) | 0, 3, and 12-14 months and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later
  The EQ-5D is a generic classification system used to characterize current health states of patients. It consists of 5 domains (mobility; self-care; usual activity; pain/discomfort; anxiety/depression) and a visual analogue scale (EQ-VAS). The domains have a scale from 1-3 and the VAS-scale from 0-100 in which higher values represent a better outcome.

SECONDARY OUTCOMES:
Change in cognitive function measured by the Neuropsychological test automated battery (CANTAB) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The investigators will use the Motor Screening Task, Reaction Time Task, Paired Associates Learning, Delayed Matching-to-Sample, Spatial Working Memory and Stop Signal Task. The higher the score on these tasks, the better the cognitive function.
Change in Depression Anxiety Stress Scale 21 (DASS-21) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The DASS-21 measures 3 related states of depression, anxiety and stress. The DASS-21 consists of 21 negative emotional symptoms and subjects will be asked to extent to which have experienced each symptom over the past week, on a 4-point severity/frequency scale. The total score will range from 0-66 in which a higher score means more susceptibility to depression.
Change in Hospital and Anxiety Scale (HADS) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The HADS will allow the investigators to measure domain-specific quality of life. This is a 14-item instrument designed to detect the presence and severity of mild degrees of mood disorder, anxiety and depression in hospital and community setting and outside. Per scale (anxiety and depression) a maximum of 21 points can be scored, in which a higher score means worse outcome.
Change in Cohen's Perceived Stress Scale (PSS) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The PSS is a measure of the degree to which situations in one's life are appraised as stressful. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Change in blood pressure after the socially evaluated cold pressure test | 0-12 months.
  The SECPT asks the participant to immerse their right hand up to and including the writs into ice water for a maximum of 3 minutes. Blood pressure will be measured before and after the test.
Change in cortisol in the saliva after the socially evaluated cold pressure test | 0-12 months.
  The SECPT asks the participant to immerse their right hand up to and including the writs into ice water for a maximum of 3 minutes. Cortisol in the saliva will be measured before and after the test.
Change in hair cortisol | 0 and 12-14 months and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Cortisol level in hair is a biomarker of chronic stress.
Change in lower extremity performance by the short physical performance battery (SPPB) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Three manoeuvres will be performed: the balance test, the gait speed test and the chair stand test. Each individual can score 0-12 points in which a higher score means a better physical performance.
Change in muscle strength by measuring handgrip strength | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Handgrip strength is measured in the dominant hand using a hydraulic grip strength dynamometer.
Change in respiratory muscle strength by measuring the inspiratory and expiratory mouth pressure | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The mouth pressure will be measured using the MicroRPM monitor.
Change in exercise performance by measuring the 6 minute walking distance | 0-12 months.
  Subjects will be instructed to walk as fast as possible for 6 minutes. The distance walked during these 6 minutes will be measured.
Change in body composition by performing Dual energy X-ray absorptiometry (DEXA-scan) | 0-12 months.
  Using the DEXA-scan three compartments of the body composition (lean mass, fat mass, bone mass) will be measured.
Change in weight | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Weight will be measured in kg.
Change in height | 0-12 months
  Height will be measured in cm.
Change in blood markers of systemic inflammation | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Markers include high-sensitive C-reactive protein, procalcitonin, interleukin-6, interleukin-8 and leucocyte levels.
Change in blood markers of nutritional status | 0-3 months; 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Markers include vitamin E, vitamin D, poly unsaturated fatty acids, amino acids (tryptophan), and homocysteine.
Change in blood markers of gut-muscle-brain cross-talk | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Markers include tryptophan, kynurenine and kynurenic acid.
Change in fatigue by using the checklist individual strength (CIS) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The CIS is a 20-item self-report questionnaire that measures several aspects of fatigue: fatigue severity, concentration, motivation and physical activity. Individual scores can range from 20-140 in which higher scores mean fatigue problems.
Change in pain using the Visual Analogue Scale (VAS) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Pain will be assessed by the VAS range from 0-100, in which a higher score means more pain experience.
Change in sleep quality by the Pittsburgh Sleep Quality Index (PSQI) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The PSQI is a self-report questionnaire to assess sleep quality. It consists of 19 individual items, creating 7 components that produce one global score (0-21, in which higher scores indicate worse sleep quality).
Change in intestinal fatty acid binding protein (blood) in rest | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  IFABP is a marker for intestinal integrity.
Change in intestinal fatty acid binding protein (blood) after the 6MWT | 0-12 months.
  IFABP is a marker for intestinal integrity.
Change in gut microbiome composition (optional) | 0, 3 and 12 months.
  Several analysis will be performed after completion of the study. The exact markers of the microbiome will be determined.

OTHER OUTCOMES:
Change in forced expiratory volume in 1 second | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Measured by spirometry within 3 previous months.
Change in forced vital capacity | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Measured by spirometry within 3 previous months.
Total lung capacity | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Measured by body plethysmography within 3 previous months
Functional residual capacity | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Measured by body plethysmography within 3 previous months
Change in diffusion capacity | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  measured within 3 previous months
Change in the global impacts of COPD on health status using the COPD assessment test (CAT) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The CAT score ranges from 0-40, in which a higher score means worse outcome.
Change in health status using the Clinical COPD questionnaire (CCQ) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The CCQ is a 10-item questionnaire and individual scores range from 0-6 in which a higher score means worse health status
Change in breathlessness using the medical research council (MRC-scale) | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  The MRC-scale ranges from 0-5 in which a higher score means more breathlessness.
Change in medication use by self-report | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  All medications used by participants will be reported to determine difference in medication use between groups.
Change in medical history will be assessed from medical records | 0-12 months; and in case of hospitalization for COPD exacerbation within one week after discharge and 4 weeks later.
  Comorbidities will be extracted from the medical history
Change in food intake | 0, 3 and 12-14 months
  3-day 24h food diary
Blood gases | in case of hospitalization for COPD exacerbation within one week after discharge
  retrieved from medical records
Type of infection | in case of hospitalization for COPD exacerbation within one week after discharge
  Viral or bacterial infection based on medical records
Number of patients died | from beginning of the study till 1 year after study completion
  from the medical records
Number of patients readmitted for a COPD exacerbation | from beginning of the study till 1 year after study completion
  from the medical records
Difference in gut microbiome composition between healthy controls and COPD patients | Baseline asssment
  To determine difference between COPD patients and healthy controls in gut microbiome composition, 30 healthy controls will sample stool at baseline which will be compared to a subgroup of 30 COPD patients.
Difference in lung function between healthy controls and COPD patients | Baseline asssment
  To ascertain that healthy controls have no obstructive lung disease, a baseline lung function measurement will be performed in the 30 healthy controls and compared to a subgroup of 30 COPD patients.
Difference in blood systemic inflammation between healthy controls and COPD patients | Baseline asssment
  To determine difference between COPD patients and healthy controls in systemic inflammation, blood samples will be obtained at baseline from 30 healthy controls and compared to a subgroup of 30 COPD patients.
Difference in food intake between healthy controls and COPD patients | Baseline asssment
  To determine difference between COPD patients and healthy controls in food intake, a 3-day 24h food diary will be obtained at baseline from 30 healthy controls and compared to a subgroup of 30 COPD patients.
Difference in medication use between healthy controls and COPD patients | Baseline asssment
  To determine difference between COPD patients and healthy controls in medication use, all medications used by the 30 healthy controls will be reported at baseline and compared to a subgroup of 30 COPD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Schols, Prof. dr., Study Director — Maastricht UMC+ / NUTRIM, Department of Respiratory Medicine
Locations (1):
- Maastricht University Medical Centre+ (MUMC+), Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
Deidentified data will only be shared based on a reasonable request.

REFERENCES:
- [Derived] van Iersel LEJ, Beijers RJHCG, Simons SO, Schuurman LT, Shetty SA, Roeselers G, van Helvoort A, Schols AMWJ, Gosker HR. Characterizing gut microbial dysbiosis and exploring the effect of prebiotic fiber supplementation in patients with COPD. Eur J Nutr. 2025 Jun 7;64(5):210. doi: 10.1007/s00394-025-03733-7. PMID 40481968
- [Derived] Beijers RJ, van Iersel LEJ, Schuurman LT, Hageman RJJ, Simons SO, van Helvoort A, Gosker HR, Schols AM. Effect of targeted nutrient supplementation on physical activity and health-related quality of life in COPD: study protocol for the randomised controlled NUTRECOVER trial. BMJ Open. 2022 Mar 16;12(3):e059252. doi: 10.1136/bmjopen-2021-059252. PMID 35296491